CLINICAL TRIAL: NCT05329363
Title: Evaluation of the Individual Early Psychoeducation Program for Schizophrenic Disorders in Inpatients: A Randomized, Multicenter Trial
Brief Title: Evaluation of the Individual Early Psychoeducation Program for Schizophrenic Disorders in Inpatients
Acronym: PEPITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DR190062
Record Dates: First submitted 2022-03-18; First posted 2022-04-15 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEPITS programme (Experimental)
  Interventions: Diagnostic Test: PEPITS Programme
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Diagnostic Test: PEPITS Programme — The programme has three main phases:
  Phase I: Introduction phase (Session 1) Phase II: Pathology and care work phase (Sessions 2 - 3 - 4) Phase III: Recovery and "stepping stone" phase (Sessions 5 - 6 - 7) The programme provides information, keys and new skills to the patient through 3 phases focusing on pathology and recovery.
  Arms: PEPITS programme
Other: Usual care — Patients will receive the same psychiatric care as the experimental group except of the PEPITS programme.
  Arms: Usual care

SUMMARY:
Schizophrenia affects about 0.7% of the population. Poor insight, which is common in this disease, linked to poor drug compliance is leads to rehospitalisation with major impact on quality of life. Indeed, many patients relapse with exacerbation of symptoms.

Psychoeducation can improve therapeutic alliance and medication compliance.

In this context, an individual psycho-education program (PEPITS) has been developed. PEPITS carried out by nurses during the initial stages of hospitalisation.

The hypothesis is that PEPITS program will decrease relapse and improve the compliance and insight and and so the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Patient with a diagnosed and reported schizophrenic disorder announced :

  * Schizophrenia
  * Schizoaffective disorder
* Or a diagnosed and reported Delusional Disorder
* Express written consent by the participant after receiving information about the study
* Be able to communicate verbally
* Participant affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient who does not speak French
* Participation in a psycho-education group in the last 2 years
* Patient under legal protection or guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evolution of insight | From inclusion (T0) up to one year (T12) after randomisation
  using the Introspection Self Assessment Questionnaire (IAQ)

SECONDARY OUTCOMES:
Evolution of patient's quality of life | From inclusion (T0) up to one year (T12) after randomisation
  using the S-QOL (Subjective - Quality of Life)
Medication compliance | From inclusion (T0) up to one year (T12) after randomisation
  by the Medication Adherence Rating Scale (MARS)
Evolution of quality of life at work | From prior to their training in the programme up to 6 months after their first inclusion
  Measured by the Quality of life at work scale (Elizur and Shye scale, validated in French by Delmas, 2001) for nurses. Score from 1 to 6 per question.
  Average of all scores.The higher the average, the higher the level of quality of life at work.
Evolution of psychological well-being at work | From prior to their training in the programme up to 6 months after their first inclusion
  Scale of psychological well-being at work (Gilbert, Dagenais-Desmarais, & Savoie, 2011) for nurses. Score from 1 to 5 per question.
  Average of all scores.The higher the average, the higher the Psychological well-being at work.
Evolution of job satisfaction | From prior to their training in the programme up to 6 months after their first inclusion
  Job satisfaction scale (Fouquereau & Rioux, 2002) for nurses. Score from 1 to 7 per question. Average of all scores. The higher the average, the higher the job satisfaction.
Evolution of sense of self-efficacy | From prior to their training in the programme up to 6 months after their first inclusion
  Self-efficacy scale (Nagels, 2008). Score from 1 to 4 per question. Average of all scores. The higher the average, the higher the sense of self-efficacy .
Evolution of commitment to work | From prior to their training in the programme up to 6 months after their first inclusion
  Work Engagement Scale (Scaufeli, Baker, & Salanova, 2006) for nurses. score from 1 to 6 per question. Average score. The higher the average, the higher the work vigour, dedication to work and absorption at work.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Serrvice de Psychiatrie, Blois
  - Service de psychiatrie, Chinon
  - Service de psychiatrie, Dreux
  - Service de psychiatrie, Fleury-les-Aubrais
  - Service de psychiatrie, La Roche-sur-Yon
  - Service de psychiatrie, Neuilly-sur-Marne
  - Service de psychiatrie, Rennes
  - Service de psychiatrie, Saint-Maurice
  - Service de psychiatrie, Sainte-Gemmes-sur-Loire
  - Service de psychiatrie, Sotteville-lès-Rouen
  - Service de psychiatrie, Tours